CLINICAL TRIAL: NCT02546518
Title: A Comparison of Surgical and a New Non-Surgical Treatment Methods for Secretory Otitis Media in Children- Hearing and Socioeconomic Aspects
Brief Title: A Comparison of Surgical and a New Non-Surgical Treatment Methods for Secretory Otitis Media in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Non-Surgical Treatment of SOM
Record Dates: First submitted 2015-09-06; First posted 2015-09-11 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Secretory Otitis Media
Keywords: Conductive hearing loss; Middle ear effusion; Middle ear pressure equalization
MeSH Terms: conditions — Otitis Media with Effusion; Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moniri Otovent (Experimental): A face mask is connected to a tube to which a coloured balloon is attached. The tube is also connected to ambu bag balloon. A safety valve is used to prevent too high air pressure. The ambu bag balloon is hidden in a green soft toy in the form of frog. The parent and the child hold the face mask against the mouth and the child blows the balloon. On need, mainly in the beginning of treatment course, the parent presses the frog's abdomen in order to fill the balloon with air. During the first week day, a low pressure balloon is used, then it is changed with a higher pressure balloon. Full compliance for the treatment is defined as 20 blows (5 minutes) in the morning and evening for one month.
  Interventions: Device: Moniri Otovent
- Tympanostomy tube in the ear drum (Active Comparator): Operation for insertion of tympanostomy tube under general anesthesia.
  Interventions: Device: Tympanostomy tube in the ear drum

INTERVENTIONS:
Device: Moniri Otovent — Please see Arm Description.
  Arms: Moniri Otovent
Device: Tympanostomy tube in the ear drum — Insertion of tympanostomy tube/Grommet in the ear drums.
  Arms: Tympanostomy tube in the ear drum

SUMMARY:
Secretory otitis media (SOM) or middle ear effusion is a common finding affecting children in the age of 4-5 years. It is usually associated with 5-15 deci Bells hearing loss. Although spontaneous resolution with normalisation of hearing is the usual outcome, this can take several months. Secretory otitis media is the most common cause of hearing impairment in the paediatric age group. When the hearing loss caused by SOM is bilateral and persists for 3-6 months or more, surgery with tympanostomy tube insertion under general anaesthesia is indicated. In Sweden, 10000 children undergo this operation annually. Although many children with unilateral or bilateral SOM improve in the summer, the problem usually recurs in the autumn or winter. The cost of SOM for the Swedish society was 600 million Swedish crowns 2005.

In two previous studies, the investigators concluded that the nonsurgical treatment method, that was developed to assist children with SOM equalising their middle ear pressure, could normalise the hearing level in 80 % of children with SOM of minimum duration of 3 months. These children avoided therefore grommet insertion.

The investigators would like to assess the effect of this new treatment method on mainly the hearing threshold of children with SOM. The investigators expect that using the new method could help children with SOM avoid operation with grommet insertion.

DETAILED DESCRIPTION:
Background:

SOM or middle ear effusion is the most common cause of hearing impairment in children. Hearing loss occurs due to the accumulation of fluid in the middle ear. In most of the cases, SOM follows acute otitis media (AOM). In cases when the SOM is bilateral and persists for more than 3-6 months, operation with grommet insertion under general anaesthesia is indicated. 10000 children with SOM are operated with grommet insertion every year in Sweden. In cases of unilateral hearing loss caused by SOM, grommet insertion is rarely indicated if the duration of symptoms is less than one year. Some patients develop persistent perforation in the eardrum after extrusion of the tympanostomy tube.

A new method of middle ear pressure equalisation has been developed at the Sahlgrenska University Hospital. 45 children in the age of 2-8 years with SOM that persisted for more than 3 months had been treated with this new method under the waiting period for grommet insertion. 80% of these children had been cured with regaining of normal hearing and avoided operation. No complication/side effects were noticed and the compliance was good.

Aim of the study:

The study aims to compare the surgical treatment with the new non surgical treatment of SOM. The effect of both treatment methods on hearing level and health economics will be assessed.

Hypothesis:

Can hearing improvement be achieved by the new non surgical treatment method of children with persistent SOM.

Material and Method:

80 children in the age of 2,5-7 years with 3-6 months duration of bilateral SOM associated with hearing loss and type B or C2 tympanogram will be offered inclusion in the study. All the patients will undergo during the first visit microscopic examination of the ears, audiogram and tympanogram. The children will be randomised thereafter into two groups. The first group is treated with the new method for one month. While the other group is operated with grommet insertion under general anesthesia. If the waiting time for the operation exceeds four weeks, the child undergo a new audiogram and tympanogram and if the results are still abnormal, the operation is performed. The second group will act as a control. Both groups undergo one month after completed treatment new examination with microscopic examination of the ears, audiogram for both groups and tympanogram for group one, due to the fact that tympanogram results are not conclusive in the presence of grommet in the ear drum.

Intervention:

The first group with verified middle ear effusion is treated with the new nonsurgical method of middle ear pressure equalisation. A face mask is connected to a tube to which a coloured balloon is attached. The tube is also connected to balloon. A safety valve is used to prevent too high air pressure. A balloon is hidden in a green soft toy in the form of frog. The parent and the child hold the face mask against the mouth and the child blows the balloon. On need, mainly in the beginning of treatment course, the parent presses the frog's abdomen in order to fill the balloon with air. During the first week, a low pressure balloon is used, then it is changed with a higher pressure balloon after one week. Full compliance for the treatment is defined as 20 blows (5 minutes) in the morning and evening for one week.

Expected results and importance:

The investigators expect that the study will show that the new treatment method of SOM, can effectively improve hearing of the affected child. This can be of great significance from medical, social and economic point of view. Hearing impairment in the paediatric age group has a great negative impact on speech development and are not only disadvantageous to the child and the parent but also for the whole society.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral secretory otitis media of 3 months duration or more
* Intact tympanic membrane bilaterally.
* Acceptable level of written and spoken swedish language skills.

Exclusion Criteria:

* Comorbidity.

Ages: 30 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hearing Level measured using age suitable audiogram. | At time of inclusion, one month, three months and six months after inclusion.
  Measuring hearing threshold using age suitable audiogram.

SECONDARY OUTCOMES:
Change from Baseline in Middle Ear Pressure measured using tympanogram. | At time of inclusion, one month, three months and six months after inclusion for the interventional group. At time of inclusion for the control group due to the fact that tympanogram is of no convenience in the presence of tympanostomy tube in the ear.
  Measuring middle ear pressure using tympanogram.
The Presence of Fluid in the Middle Ear. | At time of inclusion, one month, three months and six months after inclusion.
  Microscopic examination of the tympanic membrane to show presence of fluid in the middle ear.
Health economics measured mainly by the number of parental leave days which the parent/parents needed to take in order to look after the child. | Six months after inclusion.
Otitis Media Questionnaire-14 (OMQ-14). | At time of inclusion, three months and six months after inclusion.
  Please see Links
Number of Health Care or Hospital Visits due to Ear Associated Problems. | Six months after inclusion.
  Registration done by the parents of the number of visits to health care center or to hospital due to ear associated troubles

CONTACTS AND LOCATIONS:
Overall Officials: Hasse Ejnell, Study Director — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- See also: OMQ-14 — http://www.cmaj.ca/content/suppl/2015/07/27/cmaj.141608.DC1/141608-res-3-at.pdf